CLINICAL TRIAL: NCT06951555
Title: Controlled Study of the Effectiveness of an Individual Online (E-Health) Psychological Intervention Program for Cybersex Addiction/Online Sexual Compulsive Behavior Disorder
Brief Title: Effectiveness Study of Individual Online Treatment for Cybersex Addiction/Online Sexual Compulsive Behavior Disorder
Acronym: ADISEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P11B2015-82
Record Dates: First submitted 2025-03-07; First posted 2025-04-30 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Sexual Compulsive Behavior Disorder; Cybersex Addiction; Online Compulsive Sexual Behavior
Keywords: Cybersex addiction; psychological treatment; e-health; sexual compulsivity; effectiveness; online sex addiction
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder

STUDY DESIGN:
Intervention Model Description: Individual psychological intervention administered online with wait list control condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 12 session CBT treament
  Interventions: Behavioral: Online Individual Cognitive-Behavioral Therapy (CBT)
- Wait List Control (No Intervention): Wait list control, 3 months on wait list with no treatment

INTERVENTIONS:
Behavioral: Online Individual Cognitive-Behavioral Therapy (CBT) — 12-session individual and online CBT treatment for online sexual compulsivity/cybersex addiction
  Cognitive-behavioral psychological treatment program applied online and individually. The program consists of twelve sessions of approximately one hour's duration and weekly frequency
  1. Psychoeducational module and motivational interviewing.
  2. Environmental planning
  3. Beginning of training in emotional self-regulation techniques.
  4. Cognitive errors and cognitive discussion.
  5. Self-talk, thought traps, responsibility vs. guilt and "backpack" of coping resources.
  6. Self-esteem, stigma and life goals
  7. "Backpack" of coping resources, mindfulness and slow breathing training for anxiety
  8. Stress coping techniques
  9. Lifestyle
  10. and 11. Reduction of stimulus control and addressing previously unaddressed relevant issues.
  12. Relapse prevention
  Arms: Intervention

SUMMARY:
Cybersex addiction, understood as a subtype of Internet addiction or a manifestation of Compulsive Sexual Behavior Disorder, is a growing phenomenon. Recent studies developed by our research group have revealed that about 10% of young people in Spain could be at risk of suffering or already suffer from this problem, which can lead to consequences beyond the addiction or compulsive behavior itself, such as low self-esteem, emotional problems, sexual dysfunction, infidelity, breakups, social isolation, development of paraphilias, increase of risky sexual behavior, problems with the law, etc.. Although some studies have been carried out so far, especially on the prevalence and characterization of the sociodemographic and psychological profile of people with this disorder, psychological intervention programs for this problem have hardly been developed, and studies on the effectiveness of such programs are very scarce. Furthermore, seeking psychological help for people with this type of problem is infrequent due in part to the stigma associated with sexual addictions. In this sense, e-health approaches can reach a potential audience of users who would not access treatment if they had to physically visit a clinic. For this reason, the present project seeks to evaluate the efficacy of an online intervention aimed at the treatment of cybersex addiction or online sexual compulsive behavior disorder in the general population. For this purpose, a sample of 100 patients with a risk or pathological profile will be randomly assigned to an experimental (n=50) or control group (n=50) with similar characteristics. All of them will undergo an online assessment. The experimental group will receive an individualized online program of twelve one-hour sessions. The study will be based on an experimental design of comparison between groups (experimental-control) with pretest-posttest-follow-up evaluation at 1 month, 3 months, 6 months and 12 months, to evaluate the efficacy of the intervention. For this purpose, descriptive and differential statistical analyses (t-tests and repeated measures ANOVA), Cohen's d test for effect size and regression analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* online sexual compulsive behaviors, and may or may not also have other offline sexual compulsive behaviors
* any gender or sexual orientation
* minimum score of 9-18 points on the Internet Sex Screening Test (ISST) of Delmonico (1997) in the Spanish adaptation of Ballester, Gil, Gómez and Gil (2010)

Exclusion Criteria:

* coocurrence of psychotic symptoms, cognitive impairment, or other serious mental conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Clinical Interview for the assessment of Compulsive Sexual Behavior (SSCI-CSB) (Castro-Calvo et al., in review) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  This is a pioneering interview that allows a criterial evaluation of the patient. It asks about the different types of online and offline sexual behavior, both in terms of whether or not they are performed, as well as the percentage of sexual behavior they represent, the weekly time spent, the weekly orgasms obtained through this behavior, the discomfort it produces and the degree of control over it. From there, a series of questions related to 16 symptoms grouped around 9 criteria are developed. Then the onset, evolution, clinical course and search for therapeutic help are explored, and on the final sheet all the information can be summarized with the novelty that the diagnosis can be established according to the criteria of three classifications of three different authors (Carnes, Goodman and Kafka).
Internet Sex Screening Test (ISST) Delmonico (1997) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Spanish adaptation by Ballester, Gil, Gómez and Gil (2010). The original version includes 25 true/false items and measures online sexual behavior. Validating the original instrument with general population (through online self-administration), exploratory factor analysis revealed five factors (Delmonico and Miller, 2003): Online Sexual Compulsivity, Online Social Sexual Behavior, Online Solitary Sexual Behavior; Online Sexual Expense; and Online Sexual Behavior Interest. In addition, it includes two single-item scales. The first assesses the use of a computer outside the home for sexual purposes and the second explores access to illegal sexual material. The remaining items do not form part of any single factor. Their reliability ranged from 0.51 to 0.86. After a process of translation and adaptation of the questionnaire following the international guidelines established for this purpose (Balluerka, Gorostiaga, Alonso-Arbiol and Haranburu, 2007; Hambleton, Merenda and Spielberger, 2005
Hypersexual Behavior Inventory (Reid, Garos & Carpenter, 2011) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  This 19-item instrument with Likert-type response format (1=Never / 5=Many times) was designed to assess the three basic dimensions of hypersexuality. As noted in the introduction, the HI has been validated only in a male clinical population. In this sample, the resulting factor structure replicated the criteria under which the HI was designed. First, a factor called "Coping" (items 1, 3, 6, 8, 13, 16 and 18), which would reflect the use of sex as a means of controlling negative emotional states; secondly, another factor, "Control" (items 2, 4, 7, 10, 11, 12, 15 and 17), whose content would denote deficits in controlling sexual thoughts, impulses or behaviors; and the last factor, "Consequences" (items 5, 9, 14 and 19), which would explore persistence in sexual behavior despite the negative consequences derived. The authors obtained a high correlation between them. Reliability for each scale ranged from 0.89 to 0.95.
Sexual Compulsivity Scale (Kalichman & Rompa, 1995) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Spanish version adapted and validated for application in Spain (in preparation). This questionnaire will be used as a screening instrument from which a group of participants with sexual compulsivity problems and another group of similar number, sex, age and sexual orientation without this type of problem will be selected. The cut-off point to be used will be the same as that used by the author of the scale, the 80th percentile. Internal consistency of 0.84.
Compulsive Sexual Behavior Inventory (CSBI) (Coleman, Miner, Ohlerking & Raymond, 2001) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  28-item self-report scale that assesses the severity of symptoms of sexual compulsivity. This questionnaire is of interest because it not only includes a global measure of sexual compulsivity but also the type of compulsive paraphilic behavior (exhibitionism, sadism, phone calls, fetishism...) or non-paraphilic behavior (compulsive cruising, compulsive fixation on an unattainable partner, compulsive search for new experiences and partners, multiple sexual partners, sexual compulsivity within a specific relationship and compulsive autoeroticism).
Cognitive and Behavioral Outcomes of Sexual Behavior Scale (CBOSB) (McBride, Reece & Perera, 2006) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Following the list of consequences that may result from sexual compulsivity identified by the Society for the Advancement of the Sexual Health and classified into six domains, the authors developed this scale that records both the individual's concern about the consequences that may result from his or her sexual behavior and the fact that he or she is actually experiencing such consequences. The six domains (economic, legal, physical, psychological, spiritual and social) were identified by the National Council on Sexual Addiction and Compulsivity, NCSAC (2004) and are translated into a total of 20 items referring to cognitive aspects evaluated on a scale of 0 to 4 (never to always) and another 16 dichotomous response items that evaluate the behavioral consequences.

SECONDARY OUTCOMES:
Internet Addiction Diagnostic Questionnaire (IADQ; Young, 1998) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Questionnaire with 20 Likert-type items (rarely/occasionally/frequently/often/always). In its original version, self-administered online, it has six factors and the subscales have shown a Cronbach's alpha internal consistency between 0.54 and 0.82 (Widyanto and McMurran, 2004). Its reliability (internal consistency) in a Spanish sample of young university students is 0.910 (Salmerón, Ballester, Gómez and Gil, 2009). This questionnaire has also been recently validated by Puerta-Cortés et al. (2012) in a Colombian population.
Adapted Structured Clinical Interview for DSM, Patient Version) & SCID-II (Structured Clinical Interview for Axis II Disorders) (First, Gibbon, Spitzer, Williams & Smith) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Adaptation of SCID-P (Structured Clinical Interview for DSM, Patient version) and SCID-II (Structured Clinical Interview for Axis II Disorders) interviews (First, Gibbon, Spitzer, Williams and Smith) in a reduced version to assess psychopathological comorbidity. Especially mood disorders, anxiety disorders especially obsessive-compulsive disorder, substance use disorder, non-toxic addictions, eating disorders, personality disorders especially borderline and obsessive-compulsive disorder, sexual dysfunctions, paraphilias and other impulse control disorders.
Revised Sexual Sensation Seeking Scale (Kalichman & Rompa, 1995) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Scale evaluates one of the constructs most related to sexual compulsivity and sexual risk behaviors, sexual sensation seeking. It consists of 11 items that are answered following a 4-point Likert scale (not at all to strongly agree). Internal consistency of 0.87.
Rosenberg Self-Esteem Scale (1979) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  This questionnaire contains 10 items and provides qualitative and quantitative information on self-esteem. The high levels of validity and reliability of this scale (Cronbach's Alpha of 0.87 and test-retest reliability of 0.85) have been widely documented (Martín-Albo, Núñez, Navarro, & Grijalvo, 2007; Vázquez, Jiménez, & Vázquez-Morejón, 2004).
Hospital Anxiety and Depresión Scale (Zigmond & Snaith, 1983) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Contains 14 statements referring to symptoms of depression and anxiety, whose frequency or intensity has to be evaluated by means of a 4-point Likert scale (scores range from 0 to 3). Of the 14 items that make up the scale, 7 evaluate depression, appearing intercalary. The assessment of depression is basically limited to symptoms of anhedonia, excluding the assessment of somatic symptoms. A score above 11 points is considered as indicative of anxious or depressive symptomatology, between 8 and 10 points the symptomatology is doubtful and between 0 and 7 is considered as absence of symptomatology.
Psychological Wellbeing Scale (Ryff, 1989) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  The Ryff well-being scale assesses 6 dimensions of psychological well-being: autonomy, mastery of the environment, personal growth, positive relationships with others, purpose in life and self-acceptance. In the adaptation used, each dimension is evaluated with a thermometer, in which the patient must quantify (from 0 to 100) the extent to which they usually feel this way.
Quality of Life Index (Mezzich, Cohen & Ruiperez, 1999) | Baseline; Upon treatment completion, an average of 12 weeks; Follow-up at 1, 3, 6, and 12 months
  Assesses 10 important aspects for measuring quality of life: physical well-being, psychological well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social-emotional support, community and service support, personal fulfillment, spiritual fulfillment, global perception of quality of life.
Expectations of Change Scale (adapted from the Borkovec and Nau Inventory, 1972) | Baseline
  The original scale was designed to assess patients' credibility and expectations of improvement in therapy. In the present adaptation, after having received information about the online treatment to be received, the aim is to measure the person's expectations of change with respect to this treatment. It consists of 7 items, rated on a scale of 0 - 10 (Not at all - Very much).
Program Satisfaction Scale (adapted from the Borkovec and Nau Inventory, 1972) | Upon treatment completion, an average of 12 weeks
  After having received the treatment, it measures the person's satisfaction with the treatment in terms of liking, treatment logic, recommendation, usefulness and discomfort. It consists of seven items, rated on a scale of 0 - 10 (Not at all - Very much).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Ballester-Arnal, PhD, Principal Investigator — University Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No